CLINICAL TRIAL: NCT00002554
Title: RADIOLABELED BC8 (ANTI-CD45) ANTIBODY COMBINED WITH BUSULFAN AND CYCLOPHOSPHAMIDE AS TREATMENT FOR ACUTE MYELOGENOUS LEUKEMIA IN FIRST OR SECOND REMISSION OR UNTREATED FIRST RELAPSE FOLLOWED BY HLA-IDENTICAL RELATED MARROW TRANSPLANTATION
Brief Title: Monoclonal Antibody Followed by Bone Marrow Transplantation in Treating Patients With Acute Myelogenous Leukemia in Remission or First Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 832.00; CDR0000063421 (Registry Identifier: PDQ); NCI-V94-0393
Record Dates: First submitted 1999-11-01; First posted 2004-08-31 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Busulfan; Cyclophosphamide; Methotrexate; Radioimmunotherapy

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation
Radiation: radioimmunotherapy

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Monoclonal antibody combined with a radioactive substance and given prior to bone marrow transplantation may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of radiolabeled monoclonal antibody given prior to bone marrow transplantation in treating patients with acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the overall and disease-free survival and toxicity associated with busulfan/cyclophosphamide (BU/CTX) plus 131I-labeled BC8 antibody (131I-BC8) followed by an HLA-identical related marrow transplant in patients with acute myelogenous leukemia in first or second remission or untreated first relapse. II. Study factors that may influence the biodistribution of 131I-BC8 in this patient population, including marrow cellularity, the level of antigen expression by leukemic cells (in relapsed patients), and the degree of antigen saturation by antibody. III. Determine the efficacy of BU/CTX in patients in first remission unable to receive radiolabeled antibody, e.g., patients who are HAMA-positive, those not tolerating antibody test infusion, those with unfavorable antibody biodistribution, or those for whom antibody is unavailable.

OUTLINE: Radioimmunotherapy plus 2-Drug Cytoreductive Chemotherapy followed by Bone Marrow Transplantation with, as indicated, CNS Therapy. Iodine-131-labeled Monoclonal Antibody BC8 (anti-CD45), 131I-BC8; plus Busulfan, BU, NSC-750; Cyclophosphamide, CTX, NSC-26271; followed by Allogeneic Bone Marrow, ABM; with, as indicated, Intrathecal Methotrexate, IT MTX, NSC-740.

PROJECTED ACCRUAL: It is anticipated that 30 patients in first remission, 30 patients in untreated first relapse, and 15 patients in second remission will be accrued over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute myelogenous leukemia in first or second remission or untreated first relapse Documented CD45 expression by leukemic cells required for patients in relapse Phenotyping not required for patients in remission; such patients may have leukemia previously documented to be CD45 negative Circulating blast count less than 10,000 (control with hydroxyurea or similar agent allowed) Genotypically or phenotypically HLA-matched related marrow donor required No donors mismatched for 1 or more HLA antigens No psychologic, physiologic, or medical contraindication to donation No high risk for anesthesia because of age or medical problems No HIV seropositive donors

PATIENT CHARACTERISTICS: Age: 16 to 55 Performance status: Not specified Life expectancy: Greater than 60 days Hematopoietic: Not applicable Hepatic: Bilirubin less than 1.5 mg/dl No risk of developing veno-occlusive disease of the liver (i.e., current evidence of hepatitis as manifested by SGOT greater than 1.5 x ULN) Renal: Creatinine less than 2.0 mg/dl Other: No HIV seropositivity No major infection

PRIOR CONCURRENT THERAPY: See Disease Characteristics No prior radiotherapy to maximally tolerated levels for any normal organ

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 1993-11; Primary Completion 1999-12 (Actual); Study Completion 1999-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pagel, MD, PhD, Study Chair — Fred Hutchinson Cancer Center